CLINICAL TRIAL: NCT04665128
Title: Determining the Factors That Affects Emergency Department Visits of Hyperglycemic Patients in 30 Days.
Brief Title: Management of Hyperglycemic Patients in Emergency Medicine Department
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Derince Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Nurcihan Ulku Aytas, Emergency medicine resident, Derince Training and Research Hospital
Other Study IDs: 2020/147
Record Dates: First submitted 2020-12-07; First posted 2020-12-11 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Hyperglycemia; Diabetes Mellitus; Emergencies
MeSH Terms: conditions — Hyperglycemia; Diabetes Mellitus; Emergencies

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The main purpose of this study is how to manage hyperglycemic patients in emergency departments, to determine the conditions that require blood glucose regulation and to examine the prognosis of the patients in the next 30 days, depending on the regulation method.

DETAILED DESCRIPTION:
The study will be conducted between 15.12.2020 and 15.03.2021. Patients over the age of 18 who applied to the emergency department with any complaint and whose blood glucose level> 300 mg / dl in the examinations (as the finger tip and / or blood biochemistry examination parameter) performed in case of clinical necessity will be included in the study. Patients or their relatives (for patients who are unable to give consent) will be asked to read and sign the informed consent form if they accept it. Patients' age, gender, history, whether they are diagnosed with diabetes, medications used, vital signs, complaints of admission to the emergency room, hospitalization and definitive diagnosis will be recorded. The study form for the followed-up patients will be added to each patient's file and filled in by the physicians in the patient's follow-up.

The following parameters will be included in the work form;

1. Age of the patient
2. Gender
3. Biography
4. Presence of diabetes diagnosis, drugs used, if any
5. Other medications
6. The complaint of applying to the emergency room
7. Whether treatment for hyperglycemia is applied in the emergency department, what treatment is applied
8. How much IV fluid and / or insulin therapy is applied
9. Duration of stay in the emergency department
10. Results of routine blood tests
11. Weight
12. The trend of blood glucose levels in patients treated for hyperglycemia
13. Presence of acute complications due to hyperglycemia
14. Application and discharge BG levels
15. Whether there are classical symptoms of DM before admission to the emergency department
16. Whether hypoglycemia develops or not
17. Was medication prescribed for DM at the time of discharge?
18. Whether he was hospitalized or not. Patients will be called 30 days after leaving the emergency room (ER). Within this period, whether they applied to the emergency service again, if they did, the application complaint, the diagnosis of ER discharge, and the treatment method used will be questioned.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18, presenting to the emergency department with any complaint and with a glucose level> 300 mg / dL in blood tests will be included in the study.

Exclusion Criteria:

* Pregnant, under 18 years of age, patients who were referred to the emergency department by referral from another center, patients who received intravenous glucose treatment, patients using systemic glucocorticoids, hepatic insufficiency, renal failure, adrenal insufficiency, pancreatitis, metastatic carcinoma, patients receiving chemotherapy, patients with instability criteria will not be taken into work.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients over the age of 18, presenting to the emergency department.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2020-12-15 (Actual); Primary Completion 2021-03-15 (Estimated); Study Completion 2021-03-30 (Estimated)

PRIMARY OUTCOMES:
Reducing the glucose levels of hyperglycemic patients in the emergency department may improve clinical outcomes and have a positive effect on post-discharge prognosis. | 48 hours
  The main purpose of this study is to determine how to manage hyperglycemic patients in emergency departments, to determine the conditions that require blood glucose regulation and to examine the prognosis of the patients in the next 30 days, depending on the regulation method.

CONTACTS AND LOCATIONS:
Locations (1):
- Kocaeli Derince Training and Research Hospital, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] American Diabetes Association. 2. Classification and Diagnosis of Diabetes. Diabetes Care. 2017 Jan;40(Suppl 1):S11-S24. doi: 10.2337/dc17-S005. No abstract available. PMID 27979889
- [Background] American Diabetes Association. Diagnosis and classification of diabetes mellitus. Diabetes Care. 2014 Jan;37 Suppl 1:S81-90. doi: 10.2337/dc14-S081. No abstract available. PMID 24357215
- [Background] Fietsam R Jr, Bassett J, Glover JL. Complications of coronary artery surgery in diabetic patients. Am Surg. 1991 Sep;57(9):551-7. PMID 1928997
- [Background] Weekers F, Giulietti AP, Michalaki M, Coopmans W, Van Herck E, Mathieu C, Van den Berghe G. Metabolic, endocrine, and immune effects of stress hyperglycemia in a rabbit model of prolonged critical illness. Endocrinology. 2003 Dec;144(12):5329-38. doi: 10.1210/en.2003-0697. Epub 2003 Aug 28. PMID 12960028
- [Background] Umpierrez GE, Isaacs SD, Bazargan N, You X, Thaler LM, Kitabchi AE. Hyperglycemia: an independent marker of in-hospital mortality in patients with undiagnosed diabetes. J Clin Endocrinol Metab. 2002 Mar;87(3):978-82. doi: 10.1210/jcem.87.3.8341. PMID 11889147
- [Background] Ceriello A. Coagulation activation in diabetes mellitus: the role of hyperglycaemia and therapeutic prospects. Diabetologia. 1993 Nov;36(11):1119-25. doi: 10.1007/BF00401055. PMID 8270125
- [Background] Patel KL. Impact of tight glucose control on postoperative infection rates and wound healing in cardiac surgery patients. J Wound Ostomy Continence Nurs. 2008 Jul-Aug;35(4):397-404; quiz 405-6. doi: 10.1097/01.WON.0000326659.47637.d0. PMID 18635989
- [Background] Clement S, Braithwaite SS, Magee MF, Ahmann A, Smith EP, Schafer RG, Hirsch IB; American Diabetes Association Diabetes in Hospitals Writing Committee. Management of diabetes and hyperglycemia in hospitals. Diabetes Care. 2004 Feb;27(2):553-91. doi: 10.2337/diacare.27.2.553. No abstract available. PMID 14747243
- [Background] Gentile NT, Siren K. Glycemic control and the injured brain. Emerg Med Clin North Am. 2009 Feb;27(1):151-69, x. doi: 10.1016/j.emc.2008.08.010. PMID 19218025
- [Background] Echouffo-Tcheugui JB, Garg R. Management of Hyperglycemia and Diabetes in the Emergency Department. Curr Diab Rep. 2017 Aug;17(8):56. doi: 10.1007/s11892-017-0883-2. PMID 28646357
- [Background] Martin WG, Galligan J, Simpson S Jr, Greenaway T, Burgess J. Admission blood glucose predicts mortality and length of stay in patients admitted through the emergency department. Intern Med J. 2015 Sep;45(9):916-24. doi: 10.1111/imj.12841. PMID 26109328
- [Background] Zelihic E, Poneleit B, Siegmund T, Haller B, Sayk F, Dodt C. Hyperglycemia in emergency patients--prevalence and consequences: results of the GLUCEMERGE analysis. Eur J Emerg Med. 2015 Jun;22(3):181-7. doi: 10.1097/MEJ.0000000000000199. PMID 25222424
- [Background] Driver BE, Olives TD, Bischof JE, Salmen MR, Miner JR. Discharge Glucose Is Not Associated With Short-Term Adverse Outcomes in Emergency Department Patients With Moderate to Severe Hyperglycemia. Ann Emerg Med. 2016 Dec;68(6):697-705.e3. doi: 10.1016/j.annemergmed.2016.04.057. Epub 2016 Jun 25. PMID 27353284
- [Background] Driver BE, Olives TD, Prekker ME, Miner JR, Klein LR. The Association of Emergency Department Treatments for Hyperglycemia with Glucose Reduction and Emergency Department Length of Stay. J Emerg Med. 2017 Dec;53(6):791-797. doi: 10.1016/j.jemermed.2017.08.068. Epub 2017 Oct 6. PMID 28993036